CLINICAL TRIAL: NCT07395310
Title: A Case-Control Study on the Clinical Application Value of "Showering Cells" in the Diagnosis of Aspiration Pneumonia
Brief Title: The Clinical Application Value of "Showering Cells" in the Diagnosis of Aspiration Pneumonia
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Chief Physician, Chinese PLA General Hospital
Other Study IDs: S2025-1035-01
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia, Aspiration
Keywords: Pneumonia, Aspiration; microbiological rapid on-site evaluation (M-ROSE)
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AP Group: Adult patients with aspiration pneumonia confirmed by the composite gold standard
- Non-AP Group: Adult patients with pulmonary infection not diagnosed as aspiration pneumonia

SUMMARY:
Based on our team's previous discovery of a unique type of squamous epithelial cell in the bronchoalveolar lavage fluid (BALF) of patients with aspiration pneumonia (AP) using microbiological rapid on-site evaluation (M-ROSE) technology-characterized by its distinct morphology and absence of bacterial adhesion on the surface-which we termed "showering cells," we designed a diagnostic test case-control study. Adult patients with pulmonary infection scheduled to undergo bronchoscopy were screened and allocated into an AP group (experimental group) and a non-AP group (control group). BALF sampling and M-ROSE slide preparation were performed following a standardized protocol. Microscopic examination was conducted to detect and manually count "showering cells." Simultaneously, a committee of respiratory and critical care medicine experts determined the gold-standard diagnosis (AP or non-AP) based on composite clinical criteria.

A 2×2 contingency table was constructed to calculate sensitivity, specificity, positive/negative likelihood ratios, positive/negative predictive values along with their 95% confidence intervals, and the kappa agreement rate. A receiver operating characteristic (ROC) curve was plotted to evaluate the diagnostic performance of "showering cells" for aspiration pneumonia, from which the area under the curve (AUC) was calculated and the optimal cutoff value determined. This study aims to assess the diagnostic utility of "showering cells" and provide a novel cytomorphological tool for the diagnosis of aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 100 years, inclusive. No absolute contraindications to bronchoscopy and consent to undergo flexible bronchoscopy.

Hospitalized patients who either meet the diagnostic criteria for aspiration pneumonia or have aspiration pneumonia definitively ruled out.

AP Group：

1. Imaging Findings:Newly developed dependent infiltrates on chest CT (gravity-dependent distribution of new lung infiltrates). Specifically, in the standing/sitting position, infiltrates are predominantly seen in the basal segments of the lower lobes, especially the right lower lobe. In the supine position, infiltrates are primarily located in the posterior segment of the right upper lobe and the dorsal segment of the right lower lobe. These may be accompanied by a small amount of pleural effusion or plate-like atelectasis.
2. Clinical History Characteristics:A clear history of aspiration or the presence of at least one high-risk factor for aspiration (e.g., impaired consciousness: sedated state, post-stroke, epileptic seizure; confirmed swallowing dysfunction; gastroesophageal reflux disease; abnormal gag reflex/diminished cough reflex; poor oral hygiene: periodontitis, inadequate denture cleaning; end-stage disease: advanced dementia, malignancy, etc.).

2.Meeting 2 or more of the following 3 clinical criteria:（1）.Temperature abnormality: Fever (core temperature >38.0°C) or hypothermia (core temperature <36.0°C, more common in elderly or immunocompromised patients).(2).Respiratory symptoms: New onset or worsening of cough, production of purulent sputum (may contain food particles or unusual odor), dyspnea, chest pain, or detection of food particles/gastric contents in tracheal secretions.(3).Abnormal peripheral inflammatory markers: White blood cell count >10×10⁹/L or <4×10⁹/L, or presence of a left shift (band neutrophil proportion >5%).

Non-AP Group:

1. Imaging: Chest CT reveals newly appeared or progressive pulmonary infiltrates, consolidation, or ground-glass opacities.
2. Clinical Criteria: Meeting 2 or more of the following 3 criteria:

（1).Fever (core temperature >38.0°C) or hypothermia (core temperature <36.0°C, more common in elderly or immunocompromised patients).

(2).Respiratory symptoms: Purulent or mucopurulent sputum, possibly with blood-streaked sputum; or new/worsening cough and sputum production; or accompanied by chest pain or dyspnea.

(3).Abnormal peripheral white blood cell count: Total white blood cell count >10×10⁹/L or <4×10⁹/L, or presence of a left shift (band neutrophil proportion >5%).

3.Exclusion: Does not meet the diagnostic criteria for aspiration pneumonia.

Exclusion Criteria:

1. Younger than 18 years old or older than 100 years old.
2. Patients with absolute contraindications to performing bronchoscopy with bronchoalveolar lavage (BAL);
3. Patients who refuse to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with confirmed lung infection admitted to Chinese PLA General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
the count of "showering cells" | Day 2
  The M-ROSE examination results of BALF, specifically the count of "showering cells" across 30 high-power fields.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No